CLINICAL TRIAL: NCT04472364
Title: Impact of Blood Detection Capsule "HemoPill Acute ®" on the Time to Emergency Endoscopy in Case of Suspected Nonvariceal Upper Gastrointestinal Bleeding
Brief Title: HemoPill Acute ® in Suspected Nonvariceal Upper Gastrointestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Vivantes Netzwerk für Gesundheit GmbH (Other); University Hospital Freiburg (Other); Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Dr. med. Markus Brand, Senior Physician - Gastroenterologist, Wuerzburg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Brand_HemoPill_07_07_2020; U1111-1254-9251 (Other: WHO Universal Trail Number)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Upper Gastrointestinal Bleeding; Capsule endoscopy; Emergency endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: All participants will receive the HemoPill Acute ® capsule. In case of blood detection in the upper gi-tract (capsule positive), the endoscopy will be performed within 12 hours. If no blood is found in the upper GI tract (capsule negative), endoscopy will be performed after 48 to 96 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HemoPill (Experimental): All participants will receive the blood detection capsule HemoPill Acute ®.
  Interventions: Device: HemoPill Acute ®

INTERVENTIONS:
Device: HemoPill Acute ® — Capsule positive: Endoscopy endoscopy will be performed within 12 hours. Capsule negative: Endoscopy will be performed after 48 to 96 hours.

SUMMARY:
The study examines, whether the use of the HemoPill Acute ® capsule in case of suspected nonvariceal upper gastrointestinal bleeding can identify cases in which endoscopy can be delayed to 48-96 hours without risk to the patient.

DETAILED DESCRIPTION:
Despite a variety of scoring systems (Glasgow-Blatchford-Score, etc.) timing of endoscopy in case of suspecting nonvariceal bleeding in the upper gastrointestinal tract is still challenging.

While very early endoscopy (within 12 hours) is required in some cases, European Society of Gastrointestinal Endoscopy (ESGE) - guidelines recommend performing emergency endoscopy within 24 hours in other cases. However, a recent study (Siau et al. 2019) showed that even this time window is only kept in 59% of cases. Therefore this study examines, whether the use of the HemoPill Acute ® capsule in case of suspected nonvariceal upper gastrointestinal bleeding, can identify cases in which endoscopy can be delayed to 48-96 hours without risk to the patient.

In this study, after the routine administration of a proton pump inhibitor, hemodynamically stable emergency patients suspected of having non-variceal bleeding in the upper gastrointestinal tract receive a novel blood detection capsule (HemoPill Acute ®) for swallowing, whose result is available after 2 hours.

In case of blood detection in the upper gi-tract (capsule positive), the endoscopy will be performed within 12 hours.

If no blood is found in the upper GI tract (capsule negative), endoscopy will be performed after 48 to 96 hours, with the patient being monitored in hospital until then. In these cases, if clinical bleeding occurs before the planned endoscopy, the patient will receive an unscheduled emergency endoscopy.

Further treatment is carried out according to current clinical standards. 30 days after discharge, the patients will be asked by telephone about their further clinical course and possible complications.

The study is planned to recruit 72 participants over 48 months in several centers. If this procedure is found to be safe, the HemoPill Acute ® capsule can be used to reduce the number of emergency endoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Emergency presentation with clinical suspicion of non-variceal upper GI bleeding (e.g. haematin vomiting, melena, etc.)
* hemodynamic stable patient (heart rate <100 / min, Blood pressure sys ≥ 100mmHg)
* Emergency endoscopy indicated (modified Glasgow-Blatchford-Score ≥ 2 points)
* Administration of proton pump inhibitors possible (no allergy known)
* Good communication (without translator) with the study doctor and fulfill all requirements of the study
* Written consent after detailed information about the study

Exclusion Criteria:

* Hemodynamically unstable patients (HF> 100 / min, RR <100mmHg despite fluid administration) with indication for endoscopy within 12 hours
* Indication for endoscopy within 12 hours recommended by endoscopy call service
* Clinical suspicion of variceal bleeding of the upper GI tract (risk factors according to german guidelines: cirrhosis of the liver, splanchnic thrombosis, thrombocytopenia, known increased liver / spleen stiffness, known esophageal varices)
* Clinical suspicion of lower GI bleeding (e.g. hematochezia)
* Vomiting blood (hematemesis observed by the emergency doctor or in the clinic)
* Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Severe acute and chronic organ diseases that need treatment (e.g. kidney replacement treatment) (ASA ≥4)
* Changed anatomy of the upper GI tract (e.g. gastric resection)
* Known or suspected gastrointestinal obstructions, strictures, fistulas or known diverticula
* Dysphagia or other swallowing disorders
* Awareness restrictions that make it impossible to swallow the HemoPill Acute ® capsule on your own
* Patients with pacemakers, defibrillators, or other implantable electromedical devices
* Known allergy to parylene (capsule surface)
* Soon MRI scan planned
* Pregnancy or breastfeeding
* Mental impairment that limits the ability to meet all study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Rate of avoided emergency endoscopies (usually done within 24 hours) in case of negative HemoPill. | 48 to 96 hours after swallow the capsule
  In how many cases with a negative HaemoPill, the endoscopy interval can be extended to at least 48 hours without acute re-bleeding (confirmed in unscheduled emergency endoscopy) occurring in the meantime.
  The criteria for suspected re-bleeding (leading to an unscheduled emergency endoscopy) are: Hematemesis, again melena or hematochezia after normalized stool, tachycardia (≥110 / min) or hypotension (RRsys ≤90 mm Hg) without other explanation, decrease in the Hb value ≥2 g/dl in the course without other explanation (e.g. dilution, nosebleeds ), no increase in Hb after transfusion of erythrocyte concentrate (s) (measured after 24 hours).

SECONDARY OUTCOMES:
Rate of true positive HemoPill results leading to an emergency endoscopic intervention | 12 hours after swallow the capsule
  HemoPill positive and emergency endoscopy with active bleeding / bleeding source
Rate of false positive HemoPill results | 12 hours after swallow the capsule
  HemoPill positive and emergency endoscopy without active bleeding / bleeding source
Rate of false negative HemoPill results | 48 to 96 hours after swallow the capsule
  HemoPill negative and clinical signs of bleeding and confirmation in unscheduled emergency endoscopy
The use of the HemoPill Acute ® capsule as part of emergency care is safe and technically easy. | 30 Days after discharge
  Measurement of procedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, Prof. Dr., Principal Investigator — Universital Hospital Würzburg
Locations (4):
- Germany (4):
  - Klinikum Friedrichshain, Berlin
  - Universitästklinik Freiburg, Freiburg im Breisgau
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Universitätsklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No